CLINICAL TRIAL: NCT05330715
Title: Advanced Mobile Stroke Unit for Pre-hospital Emergency Management
Brief Title: Mobile Stroke Unit for Pre-hospital Emergency Care
Acronym: AMSU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daniel Phillips (Other Government)
Collaborators: Universität des Saarlandes (Other); East Suffolk and North Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Daniel Phillips, Clinical Lead, East of England Ambulance Service NHS Trust
Organization: East of England Ambulance Service NHS Trust (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 292195
Record Dates: First submitted 2022-03-03; First posted 2022-04-15 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Stroke, Acute; Emergencies
MeSH Terms: conditions — Stroke; Emergencies | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Mobile Stroke Unit (Other): Prehospital treatment of patients with an advanced Mobile Stroke Unit. The advanced Mobile Stroke Unit is an ambulance equipped with a computed tomography scanner, and additional diagnostic devices, such as point-of-care-laboratory and telemedicine to enable the team to diagnose and initiated specialised treatment of emergency patients at the emergency site.
  Interventions: Other: Management
- Conventional ambulance (Other): Prehospital emergency care with conventional ambulances.
  Interventions: Other: Management

INTERVENTIONS:
Other: Management — Comparison if different strategies to manage acute emergencies in the pre-hospital setting.

SUMMARY:
Emergency department overcrowding is a major challenge in medicine, leading to a delay in diagnosis and treatment for the patient due to long waiting times. This is very relevant for diseases like acute stroke and other emergencies. The Advanced Mobile Stroke Unit is an ambulance equipped with additional devices to diagnose and treat patients at the emergency site. Patients with less severe conditions can be diagnosed and safely left at home. The objectives of this project are to investigate whether the Advanced Mobile Stroke Unit compared to a normal ambulance enables more accurate triage of patients (treatment at home vs hospital vs specialist vs A&E). The Advanced Mobile Stroke Unit ambulance will be used in a random order of weeks and this will be compared to weeks with normal ambulances. The study will be carried out by the East of England Ambulance Service NHS Trust in collaboration with the East Suffolk and North Essex NHS Foundation Trust in the East of England. The project is a collaboration with Saarland University, Germany,

ELIGIBILITY:
Inclusion Criteria:

* acute emergency patients 18 years or older, who are identified via the national emergency telephone number 999 or 111with suspected severe medical emergency condition, which is categorised as: breathing problem, seizure, falls with head trauma, headache, sick person with suspected infection, stroke, unconsciousness
* calls Monday to Friday 9am to 5 pm
* written informed consent

Exclusion Criteria:

* terminally ill patients
* pregnant patients
* patients in cardiac arrest
* patients in custody of Her Majesty's prison service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 836 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-09-29 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients requiring hospital attendance within 4h of acute emergency situation | acute emergency situation (4 hours)
  Patient attendance at hospital related to the emergency call (within 4hours) will be assessed

SECONDARY OUTCOMES:
Emergency management metrics | acute emergency situation (within 4 hours after call)
  Time metrics related to the emergency call treatment (within 4 hours after call)
Clinical Outcome on day 90 | 90 days
  modified Rankin for patients with brain disease
Clinical Outcome on day 90 | 90 days
  EQ-5D5L

OTHER OUTCOMES:
Safety endpoints | 90 days
  Mortality rate within 90 days
Safety endpoints | 24 hours
  Number of patients with re-contact to EMS within 24h after emergency call
Safety endpoints | 90 days
  Number of patients with (serious) adverse events within 90 days
Health economic analysis | acute phase related to the emergency call (12 hours)
  Incremental cost-effectiveness ratio (ICER), treatment costs and health states will be evaluated for each therapy option, for the acute phase (within 12 hours)
Health economic analysis | 1 year after the acute emergency call
  Incremental cost-effectiveness ratio (ICER), treatment costs and health states will be evaluated for each therapy option after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Silke Walter, Prof, Principal Investigator — Universität des Saarlandes, EEAST
Locations (1):
- East of England Ambulance Service NHS Trust, Melbourn, United Kingdom